CLINICAL TRIAL: NCT02623868
Title: Clinical Trial to Assess the Pharmacokinetic/Pharmacodynamic Characteristics and Safety/Tolerability of CKD-519 New Formulation in Healthy Male Subjects
Brief Title: Study to Assess PK/PD Character, Safety/Tolerability of CKD-519 New Formulation in Healthy Male Subject.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 148NF15010
Record Dates: First submitted 2015-10-23; First posted 2015-12-08 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — CKD-519

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1 (Experimental): A-B-C (Drug A: CKD-519 50mg 2Tabs. /Drug B: CKD-519 100mg 1Tab. /Drug C: CKD-519 100mg 1Cap.)
  Interventions: Drug: CKD-519 50mg 2Tabs.; Drug: CKD-519 100mg 1Tab.; Drug: CKD-519 100mg 1Cap.
- Group 2 (Experimental): B-C-A (Drug A: CKD-519 50mg 2Tabs. /Drug B: CKD-519 100mg 1Tab. /Drug C: CKD-519 100mg 1Cap.)
  Interventions: Drug: CKD-519 50mg 2Tabs.; Drug: CKD-519 100mg 1Tab.; Drug: CKD-519 100mg 1Cap.
- Group 3 (Experimental): C-A-B (Drug A: CKD-519 50mg 2Tabs. /Drug B: CKD-519 100mg 1Tab. /Drug C: CKD-519 100mg 1Cap.)
  Interventions: Drug: CKD-519 50mg 2Tabs.; Drug: CKD-519 100mg 1Tab.; Drug: CKD-519 100mg 1Cap.
- Group 4 (Experimental): A-C-B (Drug A: CKD-519 50mg 2Tabs. /Drug B: CKD-519 100mg 1Tab. /Drug C: CKD-519 100mg 1Cap.)
  Interventions: Drug: CKD-519 50mg 2Tabs.; Drug: CKD-519 100mg 1Tab.; Drug: CKD-519 100mg 1Cap.
- Group 5 (Experimental): B-A-C (Drug A: CKD-519 50mg 2Tabs. /Drug B: CKD-519 100mg 1Tab. /Drug C: CKD-519 100mg 1Cap.)
  Interventions: Drug: CKD-519 50mg 2Tabs.; Drug: CKD-519 100mg 1Tab.; Drug: CKD-519 100mg 1Cap.
- Group 6 (Experimental): C-B-A (Drug A: CKD-519 50mg 2Tabs. /Drug B: CKD-519 100mg 1Tab. /Drug C: CKD-519 100mg 1Cap.)
  Interventions: Drug: CKD-519 50mg 2Tabs.; Drug: CKD-519 100mg 1Tab.; Drug: CKD-519 100mg 1Cap.

INTERVENTIONS:
Drug: CKD-519 50mg 2Tabs. — after taking Standard meal, CKD-519 50mg 2Tabs. administration.
  Other Names: Drug A
Drug: CKD-519 100mg 1Tab. — after taking Standard meal, CKD-519 100mg 1Tab. administration.
  Other Names: Drug B
Drug: CKD-519 100mg 1Cap. — after taking Standard meal, CKD-519 100mg 1Cap. administration.
  Other Names: Drug C

SUMMARY:
Study to assess the pharmacokinetic/pharmacodynamic characteristics and safety/tolerability to CKD-519 new formulation in healthy male subjects.

DETAILED DESCRIPTION:
Open-label, Randomized, 3-period, 6-sequence, crossover study

ELIGIBILITY:
Inclusion Criteria:

1. Between 20 aged and 45 aged in healthy male adult
2. Body weight ≥ 50kg and in the range of calculated BMI(Body Mass Index) 18~29kg/m2
3. Subject who sign on an informed consent form willingly
4. Necessarily he agrees that use double contraceptions and do not sperm donation until two months during clinical trials and after the final dosage of investigational products

Exclusion Criteria:

1. Clinically significant disease with cardiovascular, respiratory, hepatobiliary, nephrological, hematological, gastrointestinal, endocrine, immune, integumentary, neurologic, psychiatric system
2. Have a acute disease within 28 days before the beginning of study treatment
3. Have a disease history that can effect drug absorption, distribution, metabolism, excretion
4. Have a clinically significant chronic disease
5. Systolic blood pressure <100mmHg or >140mmHg, diastolic blood pressure<60mmHg or >90mmHg
6. Positive for serology test (HBsAg, anti-HCV Ab, anti-HIV Ab, VDRL(Venereal Disease Research Laboratories))
7. Subject treated ethical drug within 14 days before the beginning of study treatment
8. Subject treated over-the-counter or herbal medicine within 7 days before the beginning of study treatment
9. Have a clinically significant allergic disease (except for mild allergic rhinitis, allergic dermatitis with no drugs)
10. Cannot take standard Meal
11. Whole blood donation within 60 days prior to the first dosing or component blood donation within 20 days prior to the first dosing
12. Blood transfusion within 30 days
13. Taking drugs have received any other investigational drug within 90 days prior to the first dosing
14. Continuously taking caffeine(>5 cups/day), drinking alcohol(>30g/day), smoking excessive cigarettes(>10cigarettes/day)
15. Impossible on who participants in clinical trial by investigator's decision including laboratory test result or another reasone(for example, noncompliance, a disobliging manner)
16. Subject treated metabolizing enzyme inducers or inhibitors including barbiturates within 30 days

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Cmax of CKD-519 | 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 24h, 48h, 72h, 96h, 144h
Tmax of CKD-519 | 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 24h, 48h, 72h, 96h, 144h
AUClast of CKD-519 | 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 24h, 48h, 72h, 96h, 144h
AUC0-∞ of CKD-519 | 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 24h, 48h, 72h, 96h, 144h
t1/2 of CKD-519 | 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 24h, 48h, 72h, 96h, 144h
CL/F of CKD-519 | 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 24h, 48h, 72h, 96h, 144h
Vd/F of CKD-519 | 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 24h, 48h, 72h, 96h, 144h
Emax of CKD-519 CETP(Cholesteryl ester transfer protein) Activity | 0h, 1h, 2h, 4h, 6h, 8h, 10h, 12h, 16h, 24h, 48h, 72h
Tmax of CKD-519 CETP Activity | 0h, 1h, 2h, 4h, 6h, 8h, 10h, 12h, 16h, 24h, 48h, 72h
AUEC of CKD-519 CETP Activity | 0h, 1h, 2h, 4h, 6h, 8h, 10h, 12h, 16h, 24h, 48h, 72h
EC50(half maximal effective concentration ) of CKD-519 CETP Activity | 0h, 1h, 2h, 4h, 6h, 8h, 10h, 12h, 16h, 24h, 48h, 72h

CONTACTS AND LOCATIONS:
Overall Officials: Ji Young Kim, MD, PhD, Principal Investigator — Korea University
Locations (1):
- Korea university medical center, Seoul, Sungbuk-gu, South Korea